CLINICAL TRIAL: NCT06906172
Title: Effects of Plant-based Dietary Patterns on Diabetes Remission: the REmission of Diabetes Using a PlAnt-based Weight Loss InteRvention (REPAIR) Trial
Brief Title: The REmission of Diabetes Using a PlAnt-based Weight Loss InteRvention (REPAIR) Trial
Acronym: REPAIR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Unity Health Toronto (Other)
Responsible Party: Principal Investigator, Laura Chiavaroli, Assistant Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REB 24-227
Record Dates: First submitted 2025-03-17; First posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Diabetes Mellitus
Keywords: diabetes remission; weight loss; plant-based; diet; exercise; intensive lifestyle intervention; behavioural intervention; digital program
MeSH Terms: conditions — Diabetes Mellitus; Weight Loss; Motor Activity | interventions — Standard of Care

STUDY DESIGN:
Masking Description: The statistician will be masked to the treatments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- plant-based intensive lifestyle intervention (Experimental): Participants will undergo a plant-based intensive lifestyle intervention targeting weight loss with the goal of achieving diabetes remission. All antihyperglycemic and/or antihypertensive medications will be stopped at the first visit as a safety measure. The interventions will be delivered at clinic visits at 2-4week intervals over the 52-weeks.
  Interventions: Behavioral: Plant-based intensive lifestyle intervention
- standard of care (Active Comparator): Participants will continue to receive usual diabetes and obesity management with their health care provider(s) as per current Canadian clinical practice guidelines. Participants will attend clinic visits on 5 occasions over the 52-weeks.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Behavioral: Plant-based intensive lifestyle intervention — The plant-based intensive lifestyle intervention has 2 phases. The first 12-weeks is a weight loss phase consisting of a plant-based, high-plant protein energy restricted total diet replacement (TDR), psyllium-based fibre and complete multivitamin supplements, and vegetable bouillon, with the option of continuing with this phase up to week 20. The second phase is weight-loss maintenance beginning with an 8-week (weeks 12-20) stepped food reintroduction phase with partial meal replacement, progressing towards the 32-week (weeks 20-52) full food introduction phase. These phases focus on introducing a plant-based, high-plant protein, energy balanced, weight loss maintenance diet, which will be supported by a digital program. At weeks 12-28, a 16-week in-person structured exercise training program will be delivered followed by 2-weekly motivational phone calls until the 52-weeks. A 19-session, group-based, structured behavioural support program will be delivered throughout the study.
  Arms: plant-based intensive lifestyle intervention
Other: Standard of Care — Participants will continue to receive usual diabetes and obesity management as per current Canadian clinical practice guidelines. The management will continue to be delivered to participants through their family doctor, nurse practitioner, or diabetes care team with standard frequency of contact. Participants will attend clinic visits on 5 occasions (weeks 0, 12, 28, 40 and 52) and will receive motivational phone calls between visits to provide reminders regarding follow-up with their diabetes care providers.
  Arms: standard of care

SUMMARY:
The goal of this clinical trial is to learn if a plant-based intensive lifestyle intervention can achieve remission of diabetes. It will also learn if a plant-based intensive lifestyle intervention can achieve weight loss ≥15% of initial body weight.

The main questions it aims to answer are:

* What proportion of participants achieved diabetes remission (normal blood sugar for at least 3 months without medication)?
* What proportion of participants achieved ≥15% weight loss from their initial weight?
* What is the impact on weight, body composition, blood pressure, blood sugars, cholesterol and inflammation levels?

Researchers will compare the plant-based intensive lifestyle intervention to the current standard of care.

Participants will be randomly placed into one of two groups:

1. Standard of care, where they will continue their usual diabetes care with their health care providers
2. Plant-based intensive lifestyle intervention, where they will follow a diet and exercise program

Participants in the standard of care will:

* Continue with their usual diabetes care for 12 months
* Attend clinic visits on 5 occasions over the 12 months
* Allow study staff to take measurements (e.g. weight, blood pressure)
* Provide blood samples
* Track their food and exercise and complete questionnaires

Participants in the plant-based intensive lifestyle intervention will:

* Follow a plant-based low calorie diet for 3 months followed by a calorie-balanced plant-based diet for 9 months
* Participate in a 16-week exercise program
* Attend clinic visits every 2-4 weeks over the 12 months
* Allow study staff to take measurements (e.g. weight, blood pressure)
* Provide blood sample
* Track their food and exercise and complete questionnaires

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years;
* Equal number of males and females;
* Obese (body mass index [BMI] and waist circumference using sex and ethnic-specific thresholds for obesity and significant abdominal adiposity);
* Diagnosed with type 2 diabetes within the last 6 years;
* Treated by non-insulin antihyperglycemic therapy;
* Have an HbA1c 6.0-10.0%;
* Taking a stable dose of antihypertensive, antihyperglycemic, or antihyperlipidemic medications for ≥3-months, if applicable;
* Have a family physician and an Ontario Health Card;

Exclusion Criteria:

* Type 1 diabetes;
* HbA1c <6.0% or >10%;
* Recent weight loss (≥5 kg) in the last 6 months;
* Treated with diet alone;
* Treated with insulin;
* Treated with GLP-1/GIP/glucagon receptor agonist therapies;
* Treated with other anti-obesity drugs;
* Eating disorder, substance abuse disorder, serious depression, psychiatric disorder;
* Allergy or intolerance to soy;
* Allergy or intolerance to peanuts, tree nuts and seeds (all three);
* Pregnant or intending pregnancy;
* Currently breastfeeding;
* Bariatric or surgery in the last 6 months;
* Major cardiovascular event in the last 6 months;
* Kidney dysfunction;
* Unstable or severe heart failure;
* Major illness or chronic infection;
* Atherosclerotic cardiovascular disease (ASCVD);
* Chronic kidney disease (CKD);
* Treated for cancer in the last 12 months;
* Participating in another trial;
* Told by a doctor to refrain from physical activity;
* Any condition that would prevent you from following study procedures;
* Family physician does not consent to your participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2028-12-19 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Proportion achieving diabetes remission | From enrollment to the end of treatment at 52 weeks.
  Proportion achieving diabetes remission, defined as an HbA1C <6.5% for ≥3 months free of antihyperglycemic medications at 52 weeks.

SECONDARY OUTCOMES:
Key secondary: Proportion achieving ≥15% weight loss | From enrollment to the end of treatment at 52 weeks.
  Proportion achieving ≥15% weight loss from baseline at 52 weeks.
Proportion achieving ≥10% and ≥5% weight loss from baseline change | From enrollment to the end of treatment at 52 weeks
  Proportion achieving ≥10% and ≥5% weight loss from baseline at 52 weeks
Changes in measures of body composition | From enrollment to the end of treatment at 52 weeks.
  Changes in body weight
Changes in measures of body composition | From enrollment to the end of treatment at 52 weeks.
  Changes in body mass index
Changes in measures of body composition | From enrollment to the end of treatment at 52 weeks.
  Changes in waist circumference
Changes in measures of body composition | From enrollment to the end of treatment at 52 weeks.
  Changes in body fat
Changes in measures of body composition | From enrollment to the end of treatment at 52 weeks.
  Changes in lean body mass
Proportion experiencing relapse | From enrollment to the end of treatment at 52 weeks.
  Proportion experiencing relapse, defined as having achieved remission at any time during the trial but having an HbA1c ≥6.5% at 52 weeks.
Changes in functional tests | From enrollment to the end of treatment at 52 weeks.
  Changes in sit-stand chair
Changes in functional tests | From enrollment to the end of treatment at 52 weeks.
  Changes in grip test
Changes in glycemic control | From enrollment to the end of treatment at 52 weeks.
  Changes in HbA1c
Changes in glycemic control | From enrollment to the end of treatment at 52 weeks.
  Changes in fasting plasma glucose
Changes in blood lipids | From enrollment to the end of treatment at 52 weeks.
  Changes in LDL-cholesterol, non-HDL cholesterol, HDL-cholesterol, total cholesterol and triglycerides.
Changes in blood pressure | From enrollment to the end of treatment at 52 weeks.
  Changes in systolic and diastolic blood pressure.
Changes in inflammation | From enrollment to the end of treatment at 52 weeks
  Changes in c-reactive protein (CRP)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Laura Chiavaroli, MSc, PhD, Principal Investigator — University of Toronto; Dr. John L Sievenpiper, MD, PhD, FRCPC, Principal Investigator — University of Toronto, St. Michael's Hospital; Dr. David JA Jenkins, OC, MD, PhD, DSC, FRCP, FRCPSC, Principal Investigator — University of Toronto, St. Michael's Hospital; Dr. Cyril WC Kendall, PhD, Principal Investigator — University of Toronto
Locations (1):
- Unity Health Toronto (St. Michael's Hospital), Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
All outcomes listed will be shared in an anonymous/de-identified format.
Supporting Information: Study Protocol
Time Frame: IPD and supporting information will be available after the anticipated study completion date from January 2030 and will remain for 30 years until January 2060.
Access Criteria: IPD data will be accessible though the University of Toronto Dataverse (https://borealisdata.ca/dataverse/toronto). The metadata record of our dataset will be public, however access to the data will be restricted. Users will need to request access using the contact information provided in order to view and download our restricted files.